CLINICAL TRIAL: NCT05388084
Title: Peer Led Outreach to Engage Male Partners of Pregnant Women in Uganda (Okutuuka Study)
Acronym: Okutuuka
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Connie Celum, Professor: Global Health, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00014963; 1R01MH113434-01 (NIH); 1K01MH115789-01A1 (NIH)
Record Dates: First submitted 2022-05-16; First posted 2022-05-24 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Engagement, Patient; Male Peer Recruitment; HIV Testing; Linkage to Care
Keywords: Engagement, Patient; Male peer recruitment; HIV testing; PrEP; ART
MeSH Terms: conditions — Patient Participation

STUDY DESIGN:
Intervention Model Description: We will recruit pregnant women to be randomized to: 1) the intervention arm (peer father phone call) or 2) the delayed intervention arm, standard of care standard of care invitation letter to provide to their partner for fast-track HIV testing and male peer father phone calls after a 3 month delay. Women in both arms will receive an HIVST kit from the ANC clinic per standard of care guidelines. In the delayed intervention arm, men who have not HIV tested after 3 months of female partner enrollment will receive the intervention of a peer father phone call.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Male peer led intervention (Active Comparator): Male partners of women randomized to the intervention arm will receive a phone call from the male peer to encourage them to test for HIV at the clinic. Male peer fathers will offer to meet men at the clinic and guide them through the process of HIV testing. Men who are not willing/able to attend the clinic for HIV testing will be offered testing in a private and confidential location in the community; the peer male counselor meet men and offer to assist them through the process of using and interpreting an oral HIVST. Men who are not interested in testing with the peer father will be offered the HIVST kit to take home. Peer fathers will obtain men's consent to participate in the study.
  Interventions: Behavioral: Male peer engagement
- Standard of care and delayed intervention (Active Comparator): Standard of care standard of care invitation letter to provide to their partner for fast-track HIV testing and male peer father phone calls after a 3 month delay.
  Interventions: Behavioral: SOC and delayed intervention

INTERVENTIONS:
Behavioral: Male peer engagement — Male partners of women randomized to the intervention arm will receive a phone call from the male peer to encourage them to test for HIV at the clinic. Male peer fathers will offer to meet men at the clinic and guide them through the process of HIV testing. Men who are not willing/able to attend the clinic for HIV testing will be offered testing in a private and confidential location in the community; the peer male counselor meet men and offer to assist them through the process of using and interpreting an oral HIVST. Men who are not interested in testing with the peer father will be offered the HIVST kit to take home. Peer fathers will obtain men's consent to participate in the study.
  Arms: Male peer led intervention
Behavioral: SOC and delayed intervention — Females receive standard of care invitation letter to provide to their partner for fast-track HIV testing and male peer father phone calls after a 3 month delay.
  Arms: Standard of care and delayed intervention

SUMMARY:
It is critical to evaluate strategies that leverage women's engagement in antenatal care to increase male partner testing while alleviating the burden on pregnant women to encourage their male partners to HIV test. A peer-delivered status-neutral approach to male partners of pregnant women may be an innovative strategy to overcome barriers to men's reluctance to test for HIV and initiate HIV prevention or treatment services. For pregnant women living with HIV, partner testing and disclosure could facilitate women's continuation of ART post-partum, and for HIV-negative women at risk of HIV acquisition, this could facilitate women's initiation of PrEP during pregnancy. Thus, multiple public health goals could be achieved through increasing the proportion of men who know their HIV status.

DETAILED DESCRIPTION:
Overall design

This is a randomized trial of pregnant women and their male partners. The overall goal is to evaluate the impact of innovative strategies to increase male partner HIV testing and engagement in HIV care and prevention through ANC services provided to pregnant women. The intervention consists of a phone call from a trained peer father to encourage male partners of pregnant women to test for HIV. Men will first be encouraged to come to the clinic for HIV testing and counseling. Those who are not willing/able to attend the clinic will be offered the option of meeting a male counselor to receive HIV testing in a convenient location in the community. The study team will recruit pregnant women to be randomized to: 1) the intervention arm (peer father phone call) or 2) the delayed intervention arm, standard of care standard of care invitation letter to provide to their partner for fast-track HIV testing and male peer father phone calls after a 3 month delay. Women in both arms will receive an HIVST kit from the ANC clinic per standard of care guidelines. In the delayed intervention arm, men who have not HIV tested after 3 months of female partner enrollment will receive the intervention of a peer father phone call. This is being done for ethical reasons since preliminary data show phone calls from men may be effective in increasing men's HIV testing. All study outcomes will be collected by 3 months post female partner enrollment so providing the delayed intervention will not impact the study team's ability to measure the study's effectiveness. The study team will recommend that all HIV-positive participants initiate ART, and all HIV-negative participants who are eligible, initiate PrEP.

Objectives

Aim 1: To assess whether a male peer-delivered, status-neutral outreach to male partners of pregnant women increases the proportion of partners who test compared to the standard of care (invitation letters for fast-track testing and HIVST delivered by the pregnant woman).

Rationale: Innovations are needed to address the challenges associated with reaching male partners of pregnant women with HIV testing and linkage to ART or PrEP depending on their HIV serostatus.

Hypothesis: A male peer delivered, status-neutral approach to male partner engagement may overcome male partners reluctance to be tested for HIV and women's reluctance to approach their male partners about HIV testing. Approach: The investigators will randomize women 1:1 to the intervention or delayed arm and determine the proportion of male partners who test for HIV within 1 month after the female partner is randomized. The outcome will male partner testing based on male HIV testing in the two arms.

Aim 2: To determine the proportion of male partners who test HIV-negative and have an indication for PrEP who initiate PrEP and the proportion of partners who test HIV-positive who initiate ART compared to the SOC arm.

Rationale: Men who are HIV-negative are a priority for PrEP if they have a known HIV-positive partner or multiple partners, including during late pregnancy and postpartum when men are more likely to have sex with outside partners.

Hypothesis: Trained male peers will be effective in addressing men's reluctance to link to ART or PrEP and facilitating linkage to care or prevention.

Approach: Men who test for HIV through either arm will be referred for ART (if HIV-positive) or PrEP (if HIV-negative and reports multiple partners or an HIV positive partner) through the trained male peer counselor in the intervention arm or health care provider in the SOC arm. The research team will evaluate linkage to PrEP or ART among men who test for HIV, by arm.

Aim 3: To qualitatively assess acceptability of peer-delivered, status-neutral outreach to promote HIV testing among male partners of pregnant women.

Rationale: Assessment of acceptability is a key component of evaluating any novel intervention. The research team will use qualitative methods to investigate acceptability and preferences for HIV testing services among male partners of pregnant women in the cohort.

Hypothesis: A peer delivered, status-neutral approach to male partner engagement will be acceptable to recipients.

Approach: The research team will conduct individual qualitative interviews with a randomly selected subsample of 20 male partners who received peer-delivered outreach to evaluate intervention acceptability.

ELIGIBILITY:
Inclusion Criteria:

* -Age ≥18 years or if 14-17 years, qualified as emancipated minors (individuals below the age of majority who are pregnant)
* Currently pregnant
* Not currently enrolled in an HIV treatment study
* Male partner not known to be HIV-positive or has not tested in the past 3 months
* Able and willing to provide written informed consent
* Able and willing to provide adequate locator information for study retention purposes
* At low risk of intimate partner violence

For men

* Has a female partner enrolled in the Okutuuka study
* Able and willing to provide written informed consent

Exclusion Criteria:

* not meeting all of the above inclusion criteria

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Male partner HIV testing | 3 months from female partner enrollment
  The outcome for Aim 1 is the proportion of men who test for HIV in the intervention arm compared to those who test in the control arm.
  Endpoint: Site verified HIV test in a male partner of an enrolled women within three months of the women's enrollment
Linkage to PrEP | 3 months from female partner
  The outcome for Aim 2 is the proportion of male partners who test HIV-negative and have an indication for PrEP who initiate PrEP compared to the SOC arm.
Linkage to ART | 3 months from female partner
  The outcome for Aim 3 is the proportion of male partners who test HIV-positive and initiate ART compared to the SOC arm.

CONTACTS AND LOCATIONS:
Overall Officials: Connie Celum, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- Infectious Disease Institute, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Naddunga F, Bulterys MA, Nakyanzi A, Donnell D, Kyomugisha J, Birungi JE, Ssendiwala P, Nsubuga R, Muwonge TR, Musinguzi J, Peacock S, Celum CL, Mujugira A, Sharma M. Impact of male peer-led outreach on uptake of HIV testing among male partners of pregnant women in Uganda: a randomized trial. J Int AIDS Soc. 2025 Apr;28(4):e26440. doi: 10.1002/jia2.26440. PMID 40141016